## Changing Talk Online (CHATO): A Pragmatic Trial to Reduce Behavioral Symptoms in Dementia Care (Pilot)

## **Principal Investigator:**

Kristine Williams, RN, PhD, FNP-BC, FGSA, FAAN
E. Jean Hill Professor
University of Kansas School of Nursing

## Supported by:

The National Institute on Aging

**Grant number: 1R61AG061881** 

Consent - Last IRB Approval Date: August 6, 2019

We invite you to participate in a research study being conducted by investigators from the University of Kansas and the University of Iowa. The purpose of the study is to evaluate new online modules for communication training. This training has helped to improve communication in nursing homes that has reduced behavioral symptoms of residents with dementia. The goal of online modules is to improve access to this training. Evaluation will help us revise the modules to best meet the needs of direct care workers.

If you agree to participate, you will be assigned (with other participants from your nursing home) to an immediate or delayed training group. If you are in the immediate training group you will receive a URL link so you can create an account in trainingsource.org, log in, provide basic descriptive information, and complete the three modules and evaluation surveys. If you are assigned to the delayed training group, you will receive the URL link, create your account, provide descriptive information, and complete a pre-test. However, you will not complete the training modules for approximately one month when we will notify you to log in again to complete the training.

You are free to skip any questions that you prefer not to answer. It will take approximately 4 hours to complete the modules and evaluation. We will collect your name and place you work. Pre- and post-test scores and evaluation responses will only be reported for the group of participants. Your individual responses will not be reported. Data from persons completing the modules will be shared between the trainingsource.org website with the research team at the University of Kansas and the University of Iowa and may be used for future analyses.

Taking part in this research study is completely voluntary. If you do not wish to participate in this study, you don't need to do anything further. If you choose not to participate, your supervisor will not be informed. Participation rates will be shared with your nursing home as a group percentage. We appreciate your consideration.

If you have questions about the study, please contact Kristine Williams at 913-588-1673 If you have any questions about your rights as a research subject, or if you want to talk with someone who is not involved in the study, you may call the Human Subjects Committee at (913) 588-1240. You may also write the Human Subjects Committee at Mail Stop #1032, University of Kansas Medical Center, 3901 Rainbow Blvd., Kansas City, KS 66160. This study is registered on clinicaltrials.gov and can be found at: <a href="https://clinicaltrials.gov/ct2/show/NCT03849937">https://clinicaltrials.gov/ct2/show/NCT03849937</a>

Thank you very much for your consideration of this research study.